CLINICAL TRIAL: NCT05631054
Title: Establishment and Validation of a Risk Prediction Model for Long-term Low Vision After Vitrectomy in Proliferative Diabetic Retinopathy Patients
Brief Title: Establishment and Validation of a Risk Prediction Model for Long-term Low Vision After Vitrectomy in PDR Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Bojie Hu, Professor, Tianjin Medical University Eye Hospital
Other Study IDs: TianjinMUEHhbj789
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Proliferative Diabetic Retinopathy; Pars Plana Vitrectomy; Risk Prediction Model

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic retinopathy (DR) is the main cause of blindness among working-age adults in the world. Proliferative diabetic retinopathy (PDR) is the severe stage of DR, which is characterized by neovascularization of the retina. Vitreous hemorrhage and traction retinal detachment caused by PDR often require vitrectomy. The purpose of vitrectomy is to remove vitreous hemorrhage, peel off the preretinal proliferative membrane and help restore the retina. With the deepening of people's understanding of diabetes and the development and application of various hypoglycemic drugs, the life expectancy of patients with diabetes continues to prolong. Therefore, the goal of vitrectomy in patients with DR is not only to prevent blindness, but also to maintain good vision for a long time. The purpose of this study is to analyze the risk factors related to the occurrence of long-term low vision postoperatively and establish a risk prediction model, which can help patients adjust their psychological expectations reasonably and promote communication between doctors and patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and able to sign an informed consent form
* Age ≥18 years
* Documented diagnosis of diabetes mellitus (type I or type II diabetes) defined by the American Diabetes Association or World Health Organization criteria.
* Unabsorbed vitreous hemorrhage lasted for more than 2 weeks, with or without tractional retinal detachment examen by slit lamp, B-ultrasound and fundus color photography.

Exclusion Criteria:

* Patients with less than 12 months of follow-up
* Previous intraocular surgery (eg. corneal transplantation, glaucoma filtering, vitrectomy, except cataract surgery)
* Complicated with other retinal diseases
* Underwent surgery (eg. intravitreal injection, cataract surgery) of the study eye within 3 months
* Lack of medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent vitrectomy for PDR in Tianjin Medical University Eye Hospital and the follow-up period is more than 12 months. They are divided into low vision and non-low vision groups based on the BCVA at the last follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity at the last follow-up | 1 year
  Standard logarithmic visual acuity scale

SECONDARY OUTCOMES:
The occurrence of re-vitrectomy | 1 year
  The occurrence and indication of re-vitrectomy during the follow-up period
The occurrence of neovascular glaucoma | 1 year
  Non-contact computerized tonometer (CT-1, Topcon, Japan) and slit-lamp biomicroscopy
The occurrence of vitrectomy for the fellow eye | 1 year
  The occurrence of vitrectomy for the fellow eye during the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Nie Z, Xing W, Zhang X, Li X, Li W, Hu B. Association between stress hyperglycemia ratio and diabetic retinopathy progression and surgical prognosis: insights from NHANES 2005-2018 and clinical cohort study. Diabetol Metab Syndr. 2025 Jul 16;17(1):271. doi: 10.1186/s13098-025-01839-w. PMID 40671060